CLINICAL TRIAL: NCT02894411
Title: Routine Care Study Evaluating Ocular Torsion
Acronym: EXCYCLOTORSION
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: VTN_2016_18
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Superior Oblique Muscle Palsy
Keywords: MRI; Excyclotorsion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- No ocular motility disorders: Patients without ocular motility disorders, with normal orbital and brain MRI.
- superior oblique muscle palsy: Clinical features compatible with unilateral paralysis of the SO muscle Atrophy of the SO muscle on the orbital MRI without other orbital or cerebral anomaly

SUMMARY:
The paralysis of the fourth cranial nerve (paralysis IV), commonly known as the superior oblique muscle (SO) paralysis, represents half of vertical strabismus. The diagnosis of SO paralysis and of its congenital or acquired etiology, are based on a range of clinical findings. The three main clinical diagnostic elements are the hypertropia in paralyzed side which increases in adducted position, the positivity of Bielschowsky head tilt test and the twisting of the eye fundus. These criteria are always considered together and are interdependent. The diagnostic value and the sensitivity of each of these signs is not defined. Brain and orbital Magnetic Resonance Imaging (MRI) allowed a better understanding of the physiopathology of a number of oculomotor disorders.

For this reason, MRI constitute a reference for the SO palsy. The atrophy of the SO muscle is qualitatively determined by the asymmetry of muscle volume on two contiguous coronal MRI.

The diagnostic value of various clinical signs observed in SO paralysis (sensitivity, specificity) remains unknown.

ELIGIBILITY:
Inclusion Criteria:

For the subjects without oculomotor disorder

* no diplopia in different positions of gaze;
* no oculomotor disorder during the orthoptic examination (horizontal phoria <8 prism diopter, vertical phoria <4 prism diopter);
* corrected visual acuity > 8/10 on both eyes;
* binocular vision present in Lang I test (defined by 3 elements seen or appointed);
* orbital MRI: normal oculomotor muscles (including absence of atrophy of the superior oblique muscle) and lack of intra orbital expansive process;
* brain MRI: no abnormalities in the ways of oculomotor (especially no abnormalities in posterior fossa).

For the patients with SO muscle unilateral paralysis

* clinical features compatible with unilateral paralysis of the SO muscle
* muscular body atrophy of the SO on the orbital MRI without other orbital or cerebral abnormality
* binocular vision in Lang I test

Exclusion Criteria:

* high refractive error (< -6 diopter or >6 diopter);
* history or current oculomotor disorder or restrictive neurological disorder (dysthyroid orbitopathy, orbital trauma, retinal detachment surgery, paralysis oculomotor palsy other than IV);
* optic nerve head abnormalities in the fundus (edema for example)
* lack of binocular vision Lang I test;
* pregnant or breastfeeding patient
* patient under legal protection
* patient opposition to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SO muscle unilateral paralysis and patients without oculomotor disorder, matched for age.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
objective ocular torsion | baseline
  The angle of objective ocular torsion is measured on a photography of the eye fundus.

CONTACTS AND LOCATIONS:
Overall Officials: François Audren, MD, Study Director — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique A de Rothschild, Paris, France